CLINICAL TRIAL: NCT07176169
Title: Effects of Innominate Rotation Correction Compared With Sacral Torsion Correction in Patients With Sacroiliac Joint Dysfunction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/01
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-09

CONDITIONS: Sacroiliac Joint Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into two parallel groups:
  * Group A will receive Sacral Torsion Correction (via METs + Conventional Therapy)
  * Group B will receive Innominate Rotation Correction (via METs + Conventional Therapy) Both groups will undergo interventions simultaneously over a 4-week period (8 sessions total, 2 sessions/week). Outcomes will be assessed at baseline, after every second session and post-intervention, with results compared between the two groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Sacral Torsion Correction (Active Comparator): Participants allocated to this arm will receive Muscle Energy Techniques (METs) for Sacral Torsion Correction.
  Covering Patterns:
  * Left-on-Left Torsion
  * Right-on-Right Torsion
  * Left-on-Right Torsion
  * Right-on-Left Torsion
  * Bilateral Nutation
  * Bilateral Counternutation
  Each participant will undergo 8 sessions over 4 weeks (2 Sessions/week), and receive Conventional Physiotherapy
  Interventions: Procedure: Muscle Energy Technique for Sacral torsion
- Group B: Innominate Rotation Correction (Experimental): Participants allocated to this arm will receive Muscle Energy Techniques (METs) for Innominate Rotation Correction along with Conventional Treatment.
  * Anterior Rotation
  * Posterior Rotation Each participant will undergo 8 Sessions over a period of 4 weeks (2 Sessions/week).
  Interventions: Procedure: Muscle Energy Technique for Innominate rotation

INTERVENTIONS:
Procedure: Muscle Energy Technique for Sacral torsion — Conventional management including Electrotherapy by application of Thermotherapy or Cryotherapy, Transcutaneous Electrical Nerve Stimulation (TENS) for 20 minutes, Core-stabilization Exercises,
  * Clamshells
  * Four Point Kneeling
  * Bridging/Side Bridges
  * Bird-Dog Pose
  * Dead Bugs
  * Dynamic Core Stability (Unstable Surfaces) For Sacral Torsions, Six MET protocols address Forward and Backward torsions on Left and Right Oblique axis using patient generated force in Prone or Side-lying positions. Left-on-Left (LOL) Forward Torsion, Right -on-Right (ROR) Forward Torsion, Right-On-Left (ROL) Backward Torsion, Left-on-Right (LOR) Backward Torsion, Bilateral Sacral Nutation, Bilateral Sacral Counternutation
  Arms: Group A: Sacral Torsion Correction
Procedure: Muscle Energy Technique for Innominate rotation — Conventional management including Electrotherapy by application of Thermotherapy or Cryotherapy, Transcutaneous Electrical Nerve Stimulation (TENS) for 20 minutes, Core-stabilization Exercises, • Clamshells • Four Point Kneeling • Bridging/Side Bridges • Bird-Dog Pose • Dead Bugs • Dynamic Core Stability (Unstable Surfaces). Anterior Innominate Rotation and Posterior Innominate Rotation.
  Arms: Group B: Innominate Rotation Correction

SUMMARY:
The purpose of this study is to evaluate the comparative effects of Innominate Rotation Correction and Sacral Torsion Correction using Muscle Energy Techniques (METs) in patients with Sacroiliac Joint Dysfunction (SIJD). A total of 50 participants will be recruited, aged 18-50 yrs, with confirmed SIJD based on atleast 3 positive provocation tests. Participants will be randomized into two equal groups. Group A (Innominate Rotation Correction) and Group B (Sacral Torsion Correction). Both groups will receive Conventional Therapy (Thermotherapy, Electrotherapy and Core stabilization exercises).

Study variables include:

* Independent Variable: Type of MET applied (Innominate vs Sacral Torsion)
* Dependent Variables: Pain (measured by Visual Analog Scale), Functional Disability (assessed via Denver SIJ Disability Questionnaire)
* Control Variables: Age, Gender, BMI, Baseline Pain/ Disability Scores

The intervention will last 4 weeks with 8 sessions (2 sessions per week). Assessments will be conducted at baseline (Week 1, Pre-treatment) and Post every second session. Data will be analyzed to compare immediate and short-term effects of the two interventions.

This study aims to provide evidence for targeted manual therapy approaches in SIJD, potentially guiding clinicians toward the most effective technique for pain reduction and functional improvement.

DETAILED DESCRIPTION:
This Randomized Controlled Trial aims to compare the effects of Innominate Rotation Correction versus Sacral Torsion Correction using Muscle Energy Techniques (METs) in patients with Sacroiliac Joint Dysfunction (SIJD).

A Total of 50 participants will be recruited and randomized equally into two groups.

* Group A: Sacral Torsion Correction via METs
* Group B: Innominate Rotation Correction via METs

Both groups will additionally receive conventional management (TENs, Heating, Core Stabilization Exercises).

INTERVENTION SCHEDULE:

* Duration: 4 weeks
* Frequency: 2 Sessions/week
* Total Sessions: 8 Sessions per participant

Group A - Sacral Torsion Correction

* Patient Position: Side lying - depending on the torsion type
* Therapist applies downward force or guided contraction to correct torsion, with isometric contraction (3-5 sec hold), relaxation and then passive stretch.
* Each correction repeated 3-5 times.

Group B - Innominate Rotation Correction

* Patient Position: Supine
* Therapist brings limb to restrictive barrier, patient performs isometric contraction (3-5 sec) against resistance, followed by relaxation and stretch to new barrier.
* Each correction repeated 3-5 times.

ASSESSMENTS:

* Conducted at Baseline (Pre-Intervention), after every 2nd session (progress monitoring), and post-intervention (end of week 4)
* Outcomes: Pain Intensity (VAS), Functional Disability (Denver SIJD Questionnaire)

DATA ANALYSIS:

Intra-group comparisons (Pre vs Post) and Inter-group comparisons (Innominate Rotation vs Sacral Torsion) will be performed at the end of the 4-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Dysfunction based on at least 3 of the following tests

  * Distraction Test
  * Compression Test
  * Gaenslen's Test
  * Thigh Thrust Test
  * Sacral Thrust Test

    * Presence of Pain in Buttock, Posterior Pelvis, or Lower Lumbar Region for more than 2 weeks
    * Confirmed Pelvic Asymmetry through Palpation (i.e., ASIS/PSIS Landmarks, Gillet's Test)

Exclusion Criteria:

* • History of Lumbar or Pelvic Fracture, Recent Surgery, or Hip/Knee Pathology affecting Gait/Posture.

  * Pregnancy or Post-partum less than 6 months - due to Hormonal Laxity & Altered Biomechanics
  * Systemic Inflammatory conditions - Rheumatoid Arthritis, Ankylosing Spondylitis
  * Neurological Deficits - Cauda Equina Syndrome, Radiculopathy with Motor Loss
  * Ongoing Physiotherapy treatment for Low Back Pain in past 4 weeks
  * Inability/Contraindications to tolerate Manual Therapy - Osteoporosis
  * Leg Length Discrepancy - >1.5 cm or Structural Scoliosis
  * BMI > 35 (ASIA) - it may affect assessment validity due to obesity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
JOINT DISABILITY | Before and After 4 weeks.
  The Denver Sacroiliac Joint Disability Questionnaire (DSIJQ) comprises 10 items that assess various aspects of SIJ-related disability, including pain intensity, mobility, self-care, and social participation. Each item is scored on a 6-point Likert scale ranging from 0 to 5. (0 - No Disability; 5 - Unable to perform activity). To calculate the total percentage, the obtained score is divided by 50 and multiplied by 100 to calculate total percentage. Then it is compared with an Ordinal Scale grading, shown as follows:
  * 0-20% = Minimal Disability
  * 21-40% = Moderate Disability
  * 41-60% = Severe Disability
  * 61-80% = Crippled
  * 81-100% = Bed-bound or Exaggerating symptoms
JOINT PAIN | Before Treatment and After 4 weeks
  The Visual Analog Scale (VAS) is a simple patient-reported measure of current Pain Intensity.
  Scoring - Patients mark their pain on a 10-cm horizontal line, anchored by "No Pain" (0-cm) and "Worst Possible Pain" (10-cm), and the distance between 0-cm to the Point of Pain perception is marked as the recorded score (in millimeters or centimeters). High Value means Severe Pain and vice versa.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Shafay Ali, DPT, Principal Investigator — Foundation University Islamabad
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Punjab Province, Pakistan